CLINICAL TRIAL: NCT00466141
Title: Evaluation of the 2007 Shape Up RI Campaign: Study 3 Maintenance
Brief Title: Weight Maintenance Study for 2007 Shape UP RI Participants
Acronym: STOPRegain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2097-07
Record Dates: First submitted 2007-04-24; First posted 2007-04-27 (Estimated); Last update posted 2008-01-23 (Estimated); Status verified 2007-04

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Increased Exercise for weight loss maintenance
Behavioral: Daily Self-weighing for weight loss maintenance
Behavioral: Education for weight loss maintenance

SUMMARY:
This study will focus on maintenance of weight loss achieved in the 2007 Shape-Up Rhode Island(SURI)program. We plan to recruit 180 individuals who participated in SURI and lost at least 10 pounds to take part in a 4-month weight loss maintenance program when the SURI ends. Participants will be randomly assigned to one of three groups: Education, Increased Exercise, or Daily Self-Weighing.

ELIGIBILITY:
Inclusion Criteria:

1. Are 18 years or older
2. Lost 10 or more pounds during the 2007 Shape Up RI program
3. Want to learn skills to maintain your weight loss
4. Can come to the Weight Control and Diabetes Research Center located at 196 Richmond Street in the "The Jewelry District" of Providence for a baseline assessment visit in mid-May/mid-June and final assessment visit in mid-October.
5. Agree to be randomly assigned (which means you cannot choose) to one of the three weight loss maintenance interventions: General Education, Increased Physical Activity, or Self-Regulation
6. Available to take part in six 30-minute conference calls on either a Monday, Tuesday or Thursday starting at noon or 12:30pm. You will be given a toll-free call-in number so you can call from any location. The calls would be weekly for 4 weeks starting in June, and then there would be one call in mid-August and one in mid-September.

Exclusion Criteria:

1. Not 18 or more years old.
2. Did not participate in the 2007 Shape UP RI program
3. Participated in 2007 Shape Up RI but lost less than 10 pounds in the program.
4. Currently or plan to become pregnant in the next 4 months.
5. Currently participating in another weight loss or exercise study.
6. Not available to take part in six 30-minute conference calls on either a Monday, Tuesday or Thursday starting at noon or 12:30pm. The calls would be weekly for 4 weeks starting in June, and then there would be one call in mid-August and one in mid-September.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2007-06; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Wing, Ph.D, Principal Investigator — Lifespan/ The Miriam Hospital
Locations (1):
- Weight Control and Diabetes Research Center/The Miriam Hospital, Providence, Rhode Island, United States